CLINICAL TRIAL: NCT01932359
Title: Rapidly Absorbable Versus Non-absorbable Sutures for Mohs Surgery Repair on the Face: a Randomized Controlled Split-scar Study (RAVNAS)
Brief Title: Rapidly Absorbable Versus Non-absorbable Sutures for Mohs Surgery Repair on the Face: a Randomized Controlled Split-scar Study
Acronym: RAVNAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-01961
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Scars
Keywords: Scar outcome; Mohs surgery; face
MeSH Terms: conditions — Cicatrix; Facies | interventions — Nylons

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rapidly absorbable suture (Vicryl Rapide) (Active Comparator)
  Interventions: Other: rapidly absorbable suture (Vicryl Rapide)
- non-absorbable suture (Ethilon) (Active Comparator)
  Interventions: Other: non-absorbable suture (Ethilon)

INTERVENTIONS:
Other: rapidly absorbable suture (Vicryl Rapide)
  Arms: rapidly absorbable suture (Vicryl Rapide)
Other: non-absorbable suture (Ethilon)
  Arms: non-absorbable suture (Ethilon)

SUMMARY:
This study aims to compare scar outcomes between rapidly absorbable and non-absorbable sutures (stitches) for the closure of wounds after skin cancer removal on the face.

ELIGIBILITY:
Inclusion Criteria:

* Mohs surgical wound on the face
* Wound greater than or equal to 4 cm in length
* Subject is willing and capable of cooperating to the extent and degree required by the protocol and will be able to come for follow-up assessments
* Subject has read and signed Subject Information and Informed Consent Form

Exclusion Criteria:

* Surgical wound less than 4 cm in length
* Surgical site outside of face
* Subject to be be treated with radiation therapy after surgery
* Subject is not willing or able to attend for follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Stony Brook Scar Evaluation Scale (SBSES) score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Zloty, MD, Principal Investigator — University of British Columbia
Locations (1):
- Department of Dermatology and Skin Science, UBC, Vancouver General Hospital, Vancouver, British Columbia, Canada